CLINICAL TRIAL: NCT01408472
Title: CNTF Cell Implants For Glaucoma: A Phase I Study
Brief Title: NT-501 CNTF Implant for Glaucoma: Safety, Neuroprotection and Neuroenhancement
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jeffrey L Goldberg (Other)
Responsible Party: Sponsor-Investigator, Jeffrey L Goldberg, Associate Professor of Ophthalmology, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20090257
Record Dates: First submitted 2011-08-02; First posted 2011-08-03 (Estimated); Last update posted 2016-08-02 (Estimated); Status verified 2016-08

CONDITIONS: Glaucoma, Primary Open Angle
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- NT-501 CNTF Implant (Experimental): Patients will receive single NT-501 CNTF implant in one eye.
  Interventions: Drug: NT-501 CNTF Implant

INTERVENTIONS:
Drug: NT-501 CNTF Implant — Single implantation of CNTF-secreting NT-501 device into one eye

SUMMARY:
Ciliary Neurotrophic Factor (CNTF) has been demonstrated in multiple pre-clinical models to enhance survival and regeneration of retinal ganglion cells, the retinal neurons injured in diseases like glaucoma. We hypothesize that CNTF delivery to the human eye will provide neuroprotection (prevent loss of vision) and neuroenhancement (improve vision indices) in glaucoma. Patients in the trial will receive an NT-501 CNTF implant (made by Neurotech) into one eye, and will be carefully followed to evaluate safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* must understand and sign the informed consent
* must be medically able to undergo ophthalmic surgery for the NT-501 device insertion and possible removal, as well as the testing required.
* diagnosis of glaucoma characterized by (a) clinical evidence of progressive RGC dysfunction and degeneration using both visual field and at least one structural modality; (b) residual visual field preservation including best-corrected visual acuity (BCVA) better than 20/100; (c) failure to contain glaucomatous progression with maximally tolerated reduction of intraocular pressure (IOP), OR visual field defect affecting fixation, but not reducing BCVA below 20/100.

Exclusion Criteria:

* other corneal, lens, optic nerve or retinal disease causing vision loss,
* blind in one eye
* requirement of acyclovir and/or related products during study
* receiving systemic steroids or other immunosuppressive medications.
* pregnant or lactating.
* considered immunodeficient or has a known history of human immunodeficiency virus (HIV)
* on chemotherapy, or a history of malignancy, UNLESS it was treated successfully 2 years prior to inclusion in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2011-04; Primary Completion 2013-12 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Safety: Number of adverse events | 18 months
  Safety will be evaluated by counting the number of patients with adverse events, including loss of vision, visual field, or retinal/optic nerve structure, and ocular complications such as pain and inflammation.

SECONDARY OUTCOMES:
Functional Efficacy: Vision, Visual Field, Pattern Electroretinogram; Visual Field Questionnaire-25 | 18 months
Structural Efficacy: Nerve fiber layer, optic nerve topography | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey L Goldberg, MD, PhD, Principal Investigator — Bascom Palmer Eye Institute, University of Miami
Locations (1):
- Bascom Palmer Eye Institute, University of Miami, Miami, Florida, United States